CLINICAL TRIAL: NCT04515225
Title: Seroprevalence of SARS-CoV-2 Antibodies Among Adult Patients Living With HIV
Brief Title: COVID-19 Prevalence in HIV-infected Patients
Acronym: SeCoVIHA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7947
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: HIV Infections
Keywords: HIV-infection; AIDS; antiretroviral treatment; CD4 cell count; plasma HIV; RNA; SARS-CoV-2; antibodies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-infected patients: All HIV-infected patients on active follow-up, whatever clinical and biological condition, on ARV treatment or not, and whatever ARV combination
  Interventions: Other: Blood Sample

INTERVENTIONS:
Other: Blood Sample — Blood Sample

SUMMARY:
North-east area of France was hit in February 2020 by the new coronavirus disease, more severely than other French regions. Factors affecting the evolution of the disease and its severity have been quickly identified, among them figuring different kinds of immune deficiency. Even if nowadays HIV infection is usually well controlled by ARV drugs, those patients with uncontrolled viral load and/or low CD4 cell counts, remain at higher risk of severe COVID infection. In this context, the primary objective of our study is aimed at evaluating the prevalence of SARS-CoV-2 antibodies in a cohort of HIV-infected patients followed-up in an HIV-infection care center. Secondary objectives are: evaluating whether the antibodies are protective or not, the kinetic of these antibodies, and HIV associated factors with the presence of antibodies.

ELIGIBILITY:
Inclusion Criteria:

* adults (> 18 years)
* HIV-infected patients
* subjects with social insurance
* subjects able to understand study purposes, and to give a written and informed consent

Exclusion Criteria :

* subjects unable to understand informations on the study, and to provide informed consent
* subjects under guardianship or curatorship
* subjects under judicial protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients on follow-up in a single University Hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-05-03 (Estimated); Study Completion 2022-05-03 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 | From baseline to 12 months
  SARS-CoV-2 antibodies will be detected with a rapid test detecting IgG and IgM, at inclusion, and during a 6-month and a 12-month visit, in order to assess the prevalence of the virus in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No